CLINICAL TRIAL: NCT01030783
Title: A Phase 3, Randomized, Controlled, Multi-Center, Open-Label Study to Compare Tivozanib (AV-951) to Sorafenib in Subjects With Advanced Renal Cell Carcinoma (TIVO-1)
Brief Title: A Study to Compare Tivozanib (AV-951) to Sorafenib in Subjects With Advanced Renal Cell Carcinoma
Acronym: TIVO-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AV-951-09-301
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Advanced Renal Cell Carcinoma
MeSH Terms: interventions — tivozanib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tivozanib (AV-951) (Experimental)
  Interventions: Drug: tivozanib (AV-951)
- sorafenib (Active Comparator)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: tivozanib (AV-951) — Tivozanib: 1.5 mg orally once daily. Subjects will receive 1.5 mg tivozanib once daily beginning on Day 1 for 3 weeks followed by 1 week off treatment. One cycle will be defined as 4 weeks of treatment. Cycles will be repeated every 4 weeks.
  Arms: tivozanib (AV-951)
Drug: Sorafenib — Sorafenib: 400 mg orally twice daily. Subjects will receive 400 mg (2 x 200 mg tablets) sorafenib twice daily continuously, beginning on Day 1. One cycle will be defined as 4 weeks of treatment. Cycles will be repeated every 4 weeks.
  Arms: sorafenib

SUMMARY:
This is an open-label, randomized, controlled, multi-national, multi-center, parallel-arm trial comparing tivozanib to sorafenib in subjects with advanced RCC. The study is designed to compare the PFS, OS, ORR, DR, safety and tolerability, and kidney specific symptoms/health outcome measurements of tivozanib and sorafenib.

DETAILED DESCRIPTION:
This is an open-label, randomized, controlled, multi-national, multi-center, parallel-arm trial comparing tivozanib to sorafenib in subjects with advanced RCC. The study is designed to compare the PFS, OS, ORR, DR, safety and tolerability, and kidney specific symptoms/health outcome measurements of tivozanib and sorafenib.

Subjects will be randomized (1:1) to treatment with tivozanib or sorafenib and stratified by geographic region (North America/Western Europe, Central/Eastern Europe, or rest of the world); number of prior treatments (0 or 1); and number of metastatic sites/organs involved (1 or ≥ 2).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18-years of age.
2. Subjects with recurrent or metastatic RCC.
3. Subjects must have undergone prior nephrectomy (complete or partial) for excision of the primary tumor.
4. Histologically or cytologically confirmed RCC with a clear cell component (subjects with pure papillary cell tumor or other non-clear cell histologies, including collecting duct, medullary, chromophobe, mixed tumor containing predominantly sarcomatoid cells, and unclassified RCC are excluded).
5. Measurable disease per the RECIST criteria Version 1.0.
6. Treatment naïve subjects or subjects who have received no more than one prior systemic treatment (immunotherapy, including interferon-alfa or interleukin-2 based therapy, chemotherapy, hormonal therapy or an investigational agent) for metastatic RCC. Postoperative or adjuvant systemic therapy will not be counted as a prior therapy unless recurrence is detected within 6 months of completion of treatment, in which case it will be counted as a prior therapy for metastatic disease.
7. ECOG performance status of 0 or 1, and life expectancy ≥ 3 months.
8. If female and of childbearing potential, documentation of negative pregnancy test prior to enrollment.
9. Ability to give written informed consent and comply with protocol requirements.

Exclusion Criteria:

1. Any prior VEGF-directed therapy including VEGF antibody (eg, bevacizumab), VEGF receptor tyrosine kinase inhibitor (eg, sunitinib, sorafenib, axitinib, pazopanib, etc.), VEGF trap (eg, aflibercept), or any other agent or investigational agent targeting the VEGF pathway.
2. Any prior therapy with an agent targeting the mTOR pathway (eg, temsirolimus, everolimus, etc)
3. Primary CNS malignancies or CNS metastases; subjects with previously treated brain metastasis will be allowed if the brain metastasis have been stable without steroid treatment for at least 3 months following prior treatment (radiotherapy or surgery).
4. Any hematologic abnormalities (as noted in the protocol).
5. Any serum chemistry abnormalities (as noted in the protocol).
6. Significant cardiovascular disease.
7. Non-healing wound, bone fracture, or skin ulcer.
8. Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other gastrointestinal condition with increased risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to administration of first dose of study drug.
9. Serious/active infection or infection requiring parenteral antibiotics.
10. Inadequate recovery from any prior surgical procedure or major surgical procedure within 4 weeks prior to administration of first dose of study drug.
11. Significant thromboembolic or vascular disorders within 6 months prior to administration of first dose of study drug.
12. Significant bleeding disorders within 6 months prior to administration of first dose of study drug.
13. Currently active second primary malignancy, including hematologic malignancies (leukemia, lymphoma, multiple myeloma, etc.), other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer and ductal or lobular carcinoma in situ of the breast. Subjects are not considered to have a currently active malignancy if they have completed anti-cancer therapy and have been disease free for >2 years.
14. Pregnant or lactating females.
15. History of genetic or acquired immune suppression disease such as HIV; subjects on immune suppressive therapy for organ transplant.
16. Life-threatening illness or organ system dysfunction compromising safety evaluation.
17. Requirement for hemodialysis or peritoneal dialysis.
18. Inability to swallow pills, malabsorption syndrome or gastrointestinal disease that severely affects the absorption of tivozanib or sorafenib, major resection of the stomach or small bowel, or gastric bypass procedure.
19. Psychiatric disorder or altered mental status precluding informed consent or necessary testing.
20. Sexually active pre-menopausal female subjects (and female partners of male subjects) must use adequate contraceptive measures, while on study and for 50 days after the last dose of study drug. Sexually active male subjects must use adequate contraceptive measures, while on study for at least 90 days after the last dose of drug. All fertile male and female subjects and their partners must agree to use a highly effective method of contraception (including their partner). Effective birth control includes (a) IUD plus one barrier method; or (b) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm). (Note: Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are not considered effective for this study.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2009-12; Primary Completion 2012-07 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Motzer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (86):
- United States (6):
  - Site 185, Los Angeles, California
  - Site 180, Gainesville, Florida
  - Site 184, Orlando, Florida
  - Site 182, Minneapolis, Minnesota
  - Site 186, New York, New York
  - Site 187, Dallas, Texas
- Site 102, Sante Fe, Argentina
- Bulgaria (5):
  - Site 403, Plovdiv
  - Site 404, Sofia
  - Site 400, Sofia
  - Site 401, Varna
  - Site 402, Veliko Tarnovo
- Site 110, Montreal, Quebec, Canada
- Chile (3):
  - Site 121, La Reina, Santiago de Chile
  - Site 122, Santiago
  - Site 123, Temuco
- Site 411, Prague, Czechia
- France (2):
  - Site 130, Marseille
  - Site 133, Saint-Herblain
- Hungary (4):
  - Site 423, Budapest
  - Site 421, Kaposvár
  - Site 422, Pécs
  - Site 424, Szombathely
- India (12):
  - Site 157, Hyderabad, Andhra Pradesh
  - Site 190, Patna, Bihar
  - Site 156, Ahmedabad, Gujarat
  - Site 151, Nashik, Maharashtra
  - Site 153, Pune, Maharashtra
  - Site 159, Pune, Maharashtra
  - Site 191, Jaipur, Rajasthan
  - Site 155, Jaipur, Rajasthan
  - Site 152, Vellore, Tamil Nadu
  - Site 158, Lucknow, Uttar Pradesh
  - Site 150, Kolkata, West Bengal
  - Site 154, Delhi
- Italy (3):
  - Site 160, Arezzo
  - Site 161, Pavia
  - Site 162, Roma
- Poland (7):
  - Site 432, Bialystok
  - Site 434, Bydgoszcz
  - Site 431, Gdansk
  - Site 435, Olsztyn
  - Site 433, Poznan
  - Site 430, Warsaw
  - Site 436, Warsaw
- Romania (5):
  - Site 444, Brasov
  - Site 441, Bucharest
  - Site 440, Bucharest
  - Site 443, Bucharest
  - Site 442, Timișoara
- Russia (19):
  - Site 459, Ufa, Bashkortostan Republic
  - Site 451, Chelyabinsk
  - Site 452, Kazan'
  - Site 454, Moscow
  - Site 453, Moscow
  - Site 458, Moscow
  - Site 460, Moscow
  - Site 461, Moscow
  - Site 462, Moscow
  - Site 450, Nizhny Novgorod
  - Site 456, Obninsk
  - Site 467, Omsk
  - Site 463, Pyatigorsk
  - Site 457, Rostov-on-Don
  - Site 466, Saint Petersburg
  - Site 465, Saint Petersburg
  - Site 464, Yaroslavi
  - Site 455, Yekaterinburg
  - Site 468, Yoshkar-Ola
- Serbia (5):
  - Site 480, Belgrade
  - Site 481, Belgrade
  - Site 482, Belgrade
  - Site 484, Kamenitz
  - Site 483, Niš
- Ukraine (9):
  - Site 491, Chernihiv
  - Site 492, Dniproperovsk
  - Site 498, Dnipropetrovsk
  - Site 493, Donetsk
  - Site 496, Donetsk
  - Site 490, Ivano-Frankivsk
  - Site 494, Kharkiv
  - Site 497, Uzhhorod
  - Site 495, Zaporizhia
- United Kingdom (3):
  - Site 170, Cambridge
  - Site 173, Ipswich
  - Site 172, Leicester

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- See also: Related Info — http://www.aveopharma.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tivozanib (AV-951) | Sorafenib
Started | 260 | 257
Completed | 211 | 231
Not Completed | 49 | 26

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Tivozanib (AV-951) | Sorafenib | Total
Number analyzed (Participants) | 260 | 257 | 517
Age, Continuous [Median (Full Range); unit: Years] | 59 [23 to 83] | 59 [23 to 85] | 59 [23 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 68 | 143
  Male | 185 | 189 | 374

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) of Subjects With Advanced Renal Cell Cancer (RCC) Randomized to Treatment With Tivozanib or Sorafenib
Description: Progression-Free Survival (PFS) is defined as the time from randomization to first documentation of objective tumor progression (progressive disease) or death due to any reasons whichever comes first. Disease progression per RECIST 1.0 criteria is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first. Disease progression was assessed every 8 weeks.
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tivozanib (AV-951) | Sorafenib
Number analyzed (Participants) | 260 | 257
Months | 11.9 [9.3 to 14.7] | 9.1 [7.3 to 9.5]

2. Secondary Outcome: Overall Survival (OS) of Subjects Randomized to Treatment With Tivozanib or Sorafenib
Description: Overall survival (OS) is defined as the time from the date of randomization to date of death due to any cause. In the absence of confirmation of death, survival time will be censored at the last date the subject is known to be alive. Subjects lacking data beyond randomization will have their survival times censored on the date of randomization.
Time Frame: Date of randomization to date of death
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tivozanib (AV-951) | Sorafenib
Number analyzed (Participants) | 260 | 257
Months | 28.2 [22.5 to 33.0] | 30.8 [28.4 to 33.3]

3. Secondary Outcome: Objective Response Rate (ORR) of Subjects Randomized to Treatment With Tivozanib or Sorafenib
Description: Objective response rate (ORR) is defined as the percentage of subjects who have at least a 30% reduction in the sum of diameters per RECIST (Version 1.0).
Time Frame: Every 8 weeks from date of randomization until disease progression
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tivozanib (AV-951) | Sorafenib
Number analyzed (Participants) | 260 | 257
percentage of participants | 33.1 [27.4 to 39.2] | 23.3 [18.3 to 29.0]

4. Secondary Outcome: Duration of Response (DR) of Subjects Randomized to Treatment With Tivozanib or Sorafenib
Description: Duration of response (DR) is defined as the time from the first documentation of objective tumor response to the first documentation of tumor progression per RECIST 1.0 or to death due to any cause.
Time Frame: Assessed every 8 weeks from date of randomization until date of progression
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tivozanib (AV-951) | Sorafenib
Number analyzed (Participants) | 86 | 58
Months | 15.0 [12.9 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event. | 12.9 [11.0 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event.

5. Secondary Outcome: Safety and Tolerability of Tivozanib and Sorafenib
Description: Dose reductions and interruptions were allowed for subjects taking tivozanib or sorafenib. Any modification of study drug administration, and the reason for such action, was clearly noted on the subject's eCRF.
Time Frame: From start of treatment therapy to completion of treatment therapy, an average of 11 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Tivozanib (AV-951) | Sorafenib
Number analyzed (Participants) | 259 | 257
Participants
  Reasons for Dose Interruptions - Adverse Event | 50 | 92
  Reasons for Dose Reductions - Adverse Event | 36 | 111

6. Secondary Outcome: To Compare Kidney-specific Symptoms and Health Outcome Measurements in Subjects Randomized to Treatment With Tivozanib or Sorafenib
Description: The Disease Related Symptom Scale of the Functional Assessment of Cancer Therapy - Advanced Kidney Cancer Symptom Index (FKSI-DRS) measured kidney specific symptoms on a 0-36 scale, with lower scores corresponding to worse overall QOL and higher scores corresponding to better overall QOL. The Functional Assessment of Cancer Therapy-General (FACT-G) measured general wellbeing scored on a 0-108 scale, with lower scores corresponding to worse overall QOL and higher scores corresponding to better overall QOL. The European Quality of Life-5 Dimensions (EQ-5D) measured patient health related quality of life scored on a 0-1 scale, with 0 being worse health state and 1 being perfect health state. The European Quality of Life-5 Dimensions Visual Analog Scales (EQ-5D VAS) measured patient health related quality of life on a visual analog scale from 0 to 100, with 0 being the worst and 100 being the best. These scales were self-administered by patients at the start of the visit.
Time Frame: At Day 1 of each 28 day cycle throughout the course of the study, for an average of 11 months per subject
Population: ITT Population, excluding questionnaires that were not analyzable
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tivozanib (AV-951) | Sorafenib
Number analyzed (Participants) | 257 | 250
Score on a scale
  FACT-G Total Score: number analyzed (Participants) | 257 | 248
  FACT-G Total Score | 74.16 (0.785) | 73.05 (0.802)
  FKSI-DRS Score: number analyzed (Participants) | 256 | 248
  FKSI-DRS Score | 28.71 (0.227) | 28.58 (0.233)
  EQ-5D Weighted Health State Index: number analyzed (Participants) | 256 | 250
  EQ-5D Weighted Health State Index | 0.67 (0.014) | 0.66 (0.014)
  EQ-5D VAS | 71.50 (0.826) | 68.49 (0.841)

7. Secondary Outcome: Pharmacokinetics (Serum Concentrations) of Tivozanib
Description: Samples for tivozanib serum concentrations will be collected at the following time points: Cycle 1, Day 1 (prior to dosing), Cycle 1, Day 15 (prior to dosing), Cycle 2, Day 1 (prior to dosing), and Cycle 2, Day 22-28. The serum concentrations of tivozanib were tabulated for individual subjects and summarized by nominal time using standard descriptive statistics (concentrations presented in ng/mL).
Time Frame: Cycle 1, Day 1 (prior to dosing), Cycle 1, Day 15 (prior to dosing), Cycle 2, Day 1 (prior to dosing), and Cycle 2, Day 22-28
Population: All patients who had taken at least 1 dose of tivozanib and who had at least one measurable concentration value.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Tivozanib (AV-951)
Number analyzed (Participants) | 254
ng/mL
  Cycle 1, Day 1: number analyzed (Participants) | 249
  Cycle 1, Day 1 | 0 [0.0 to 0.0]
  Cycle 1, Day 15: number analyzed (Participants) | 250
  Cycle 1, Day 15 | 69.05 [65.0 to 73.1]
  Cycle 2, Day 1 | 30.87 [28.0 to 33.7]
  Cycle 2, Day 22-28: number analyzed (Participants) | 244
  Cycle 2, Day 22-28 | 54.37 [49.8 to 59.0]

ADVERSE EVENTS:
Time Frame: From first dose to last dose plus 30 days, approximately 1 year on average
Description: Safety Population
Arm/Group | Tivozanib (AV-951) | Sorafenib
Serious Adverse Events (participants affected / at risk) | 74/259 | 56/257
Other Adverse Events (participants affected / at risk) | 238/259 | 249/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tivozanib (AV-951) (N=259) | Sorafenib (N=257)
Cerebrovascular accident (Nervous system disorders) | 4 | 3
Ischaemic stroke (Nervous system disorders) | 3 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 2
Acute myocardial infarction (Cardiac disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 2 | 4
Fatigue (General disorders) | 3 | 1
Death (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 4 | 4
Hypertension (Vascular disorders) | 3 | 2
Pneumonia (Infections and infestations) | 1 | 3
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 3
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Periproctitis (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Salivary gland mass (Gastrointestinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Abscess soft tissue (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fluid collection (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Amylase increased (Investigations) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tivozanib (AV-951) (N=259) | Sorafenib (N=257)
Hypertension (Vascular disorders) | 116 | 91
Diarrhoea (Gastrointestinal disorders) | 63 | 85
Nausea (Gastrointestinal disorders) | 34 | 19
Stomatitis (Gastrointestinal disorders) | 30 | 23
Vomiting (Gastrointestinal disorders) | 20 | 12
Abdominal pain upper (Gastrointestinal disorders) | 18 | 17
Abdominal pain (Gastrointestinal disorders) | 16 | 10
Constipation (Gastrointestinal disorders) | 12 | 13
Fatigue (General disorders) | 53 | 41
Asthenia (General disorders) | 44 | 44
Pyrexia (General disorders) | 11 | 13
Weight decreased (Investigations) | 49 | 54
Blood thyroid stimulating hormone increased (Investigations) | 14 | 6
Lipase increased (Investigations) | 12 | 24
Blood phosphorus decreased (Investigations) | 5 | 16
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 55 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 38 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 6
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 36 | 139
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 55
Rash erythematous (Skin and subcutaneous tissue disorders) | 6 | 16
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 13
Rash papular (Skin and subcutaneous tissue disorders) | 3 | 16
Headache (Nervous system disorders) | 23 | 11
Decreased appetite (Metabolism and nutrition disorders) | 28 | 24
Proteinuria (Renal and urinary disorders) | 24 | 21
Anaemia (Blood and lymphatic system disorders) | 15 | 15
Hypothyroidism (Endocrine disorders) | 14 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No